CLINICAL TRIAL: NCT06695897
Title: Prospective, Non-interventional Observational Study to Characterize Dupilumab in the Long-term Management of Eosinophilic Esophagitis, Safety and Patient Reported Outcomes (Quality of Life) in Clinical Routine
Brief Title: A Non-interventional Observational Study to Assess Long-term Efficacy and Safety of Dupilumab for the Treatment of Patients (>= 12 Years) With Eosinophilic Esophagitis Under Real-world-conditions in Germany
Acronym: ProMEAL
Status: Recruiting | Type: Observational
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: OBS18402; U1111-1306-7545 (Registry Identifier: ICTRP)
Record Dates: First submitted 2024-11-15; First posted 2024-11-19 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Eosinophilic Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis | interventions — dupilumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Dupilumab arm: Patients who receive dupilumab for eosinophilic esophagitis (EoE) treatment in a real-world setting in Germany
  Interventions: Drug: Dupilumab

INTERVENTIONS:
Drug: Dupilumab — This study will not administer any treatment, only observe the treatment as prescribed in real-world clinical practice.

SUMMARY:
This is a longitudinal, observational non-interventional study (NIS) designed to characterize the patient population who receives dupilumab for eosinophilic esophagitis (EoE) treatment in a real-world setting in Germany with respect to their medical history, socio-demographic and disease characteristics, comorbidities (including type 2 inflammatory and atopic conditions), concomitant therapies and prior EoE treatments. Furthermore, this NIS aims to describe the long-term effectiveness of dupilumab for the treatment of EoE as assessed by the treating physician and reported by the patient, and its effect on health-related quality of life (HRQoL) during an individual observational period of two years. In addition, data on real-world use patterns and long-term safety data of dupilumab treatment for EoE will be collected.

DETAILED DESCRIPTION:
The study duration for each participant is planned to be 2 years. Total study duration is approximately 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with EoE who are inadequately controlled by, are intolerant to, or who are not candidates for conventional medicinal therapy
* Patients for whom the treating physician has decided to initiate new treatment with dupilumab for EoE according to EU-SmPC independently from entry in study or for whom treatment with dupilumab for EoE according to EU-SmPC has been started within the last 7 days. The decision to initiate dupilumab treatment is made by the treating physician and the patient according to the patient´s medical need and to the standard of best medical practice. This decision is made independently and before inclusion in this NIS.
* ≥ 12 years of age at baseline visit
* ≥ 40 kg bodyweight
* Voluntary study participation and signed written informed consent by patient and parent(s)/guardian(s), if applicable

Exclusion Criteria:

* Patients who have a contraindication to dupilumab according to the current EU-SmPC.
* Patients who have been treated with dupilumab for more than 7 days
* Any acute or chronic condition that, in the treating physician´s opinion, would limit the patient´s ability to complete questionnaires or to participate in this study or impact the interpretation of the results.
* Participation in an ongoing interventional or observational study that might, in the treating physician´s opinion, influence the assessments for the current study (parallel inclusion in another Sanofi-independent registry might be possible if the patient gives consent)

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients suffering from EoE, ≥ 12 years of age with at least 40 kg bodyweight who are planned to be initiated with dupilumab for the treatment of EoE according to the prescribing information, i.e., the current Summary of Product Characteristics approved in the European Union (EU-SmPC).
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2029-05-29 (Estimated)

PRIMARY OUTCOMES:
Descriptive statistical analysis of medical history characteristics | At baseline
Descriptive statistical analysis of socio-demographic characteristics | At baseline
Descriptive statistical analysis of disease characteristics | At baseline

SECONDARY OUTCOMES:
Absolut change from baseline in endoscopic reference score (EREFS) | After 3, 6 (optional), 12 and 24 months of dupilumab treatment
  Absolut change from baseline in EREFS (including inflammatory and fibrostenotic subscore)
Proportion of patients with eosinophils per high power field (EOS/hpf) < 15 in esophageal biopsies | After 3, 6 (optional), 12 and 24 months of dupilumab treatment
Change in clinical symptoms from baseline | From baseline until 1, 3, 6, 9, 12, 18 and 24 months of dupilumab treatment
  Change in clinical symptoms (as assessed in clinical practice) from baseline
Behavioral changes regarding food intake from baseline | From baseline until 1, 3, 6, 9, 12, 18 and 24 months of dupilumab treatment
  Behavioral changes regarding food intake (as reported by the patient)
Absolute change from baseline in Dysphagia Numerical Rating Scale (NRS) | After 1, 3, 6, 9, 12, 18 and 24 months of dupilumab treatment
  Scale from 0 (no trouble to swallow) - 10 (maximum trouble to swallow)
Absolute change from baseline in Hospital Anxiety and Depression Scale (HADS) | After 1, 3, 6, 9, 12, 18 and 24 months of dupilumab treatment
Absolute change from baseline Pediatric Eosinophilic Esophagitis Symptom Scores (PEESS v2.0) | After 1, 3, 6, 9, 12, 18 and 24 months of dupilumab treatment
Absolute change from baseline Pediatric Quality of Life Inventory (PEDS-QL) | After 1, 3, 6, 9, 12, 18 and 24 months of dupilumab treatment
Number of hospitalizations due to EoE | During the last 12 months before baseline and after 12 and 24 months of dupilumab treatment
Number of sick leave days at work due to EoE | During the last 12 months before baseline and after 12 and 24 months of dupilumab treatment
Reason(s) for initiation of dupilumab treatment | At baseline
Descriptive statistical analysis of details on dupilumab treatment | Throughout the study, for approximately 24 months after dupilumab treatment
  Descriptive analysis: form of administration, location of administration
Analysis of treatment emergent adverse events (TEAEs) | Throughout the study, for approximately 24 months after initiation of dupilumab treatment
  Quantity of treatment emergent adverse events, quantity of TEAE that lead to ending of therapy, collection of type of TEAE

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number: 0000001, Dachau, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org